CLINICAL TRIAL: NCT02145065
Title: Prospective, Pivotal, First - in Man Clinical Trial of the Safety and Efficacy of a Novel Microcrystalline Paclitaxel Coated Balloon for Treatment of Femoropopliteal Artery Disease
Brief Title: First-in-man Evaluation of a Novel, Microcrystalline Paclitaxel Coated Balloon for Treatment of Femoropopliteal Artery Disease (PAX-r)
Acronym: PAX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Balton Sp.zo.o. (Industry)
Collaborators: American Heart of Poland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PAX-0314
Record Dates: First submitted 2014-05-20; First posted 2014-05-22 (Estimated); Last update posted 2018-08-07 (Actual); Status verified 2018-08

CONDITIONS: Peripheral Artery Disease; Femoropopliteal Artery Disease
Keywords: paclitaxel coated balloon; restenosis; Femoropopliteal artery disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Plain Balloon Angioplasty (Active Comparator): Plain Balloon Angioplasty
  Interventions: Device: Plain balloon angioplasty, uncoated balloon (Neptun, Balton, Poland)
- microcrystalline Paclitaxel Coated Balloon (PAK) (Experimental): plain balloon angioplasty followed by mcPCB dilation
  Interventions: Drug: Local drug delivery via microcrystalline paclitaxel balloon coating (PAK,Balton, Poland)

INTERVENTIONS:
Drug: Local drug delivery via microcrystalline paclitaxel balloon coating (PAK,Balton, Poland)
  Arms: microcrystalline Paclitaxel Coated Balloon (PAK)
Device: Plain balloon angioplasty, uncoated balloon (Neptun, Balton, Poland)
  Arms: Plain Balloon Angioplasty

SUMMARY:
The purpose of this pivotal, first in man study will be to evaluate safety and efficacy of the novel, microcrystalline paclitaxel coated balloon (mcPCB, PAK, Balton) in the treatment of femoropopliteal artery disease.

DETAILED DESCRIPTION:
Although clinically effective, the manufacturing process of first generation PCB coatings contributed to inconsistent drug concentrations, particulate formations on the balloon surface and their shedding during the interventional procedures. As a consequence developments of new PCB coatings have been proposed to address consistency, uniformity, small particle drug coverage, which may potentially contribute to improved vessel healing profile and improved clinical outcomes. Nevertheless, data on the safety and efficacy of this novel coating developments in the clinical setting remain limited. Previously in the experimental model, the investigators reported that delivery of paclitaxel via a novel mcPCB resulted in low long-term tissue retention of paclitaxel, however displayed reduced neointimal proliferation and favorable healing profile. Therefore in current clinical trial the investigators will address the feasibility and safety of the mcPCB (PAK, Balton) in the treatment of femoropopliteal restenotic disease in a prospective, randomized manner when compared to plain balloon angioplasty (PBA). The efficacy analysis will be observational and evaluated post-hoc, with no prespecified criteria.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 y.o.
* Claudication in Rutherford Class 1-5,
* Lesion in the femoropopliteal artery defined as >50% and < 99% diameter stenosis with length of up to 10 cm in vessel diameter of 3-7 mm
* Chronic total occlusions of length less than 100 mm
* Ability to cross the lesions with a guidewire.

Exclusion Criteria:

* Critical acute or chronic limb ischemia
* Acute coronary syndrome
* Chronic kidney disease stage III-V
* Restenotic lesion
* Femoropopliteal graft
* Known allergy to clopidogrel or aspirin
* History of stroke within past 6 months
* Age > 80 y.o.
* Life expectancy < 2 years

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2014-09; Primary Completion 2017-09 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Angiographic late lumen loss | 6 months

SECONDARY OUTCOMES:
Safety - Device related adverse events | 30 days, 6 months
Critical limb ischemia | 30 days, 6 months
Device Success | at procedure
  Successful delivery and deployment of the first inserted study device (in overlapping setting a successful delivery and deployment of the first and second study device) at the intended target lesion and successful withdrawal of the study device with attainment of final residual stenosis of less than 30% of the target lesion by quantitative vessel angiography (QVA).
Target Lesion Revascularization | 6, 12, 24 months
Target vessel revascularization | 6, 12, 24 months
Primary patency of treated segment | 6, 12, 24 months
Treated limb amputation | 30 days, 6 months

OTHER OUTCOMES:
Change in ankle-brachial index | pre-procedure, 3,6 and 12 months
Change in Walking Impairment Questionnaire (WIQ) | pre procedure, 3, 6 and 12 months
Flow velocity in doppler ultrasonography | 3, 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Przemysław Nowakowski, M.D., PhD, Principal Investigator — American Heart of Poland, Katowice, Poland; Piotr P Buszman, M.D., PhD, Principal Investigator — American Heart of Poland, Katowice, Poland
Locations (1):
- Lesser-Poland Cardiovascular Center of American Heart of Poland, Chrzanów, Poland

REFERENCES:
- [Background] Buszman PP, Milewski K, Zurakowski A, Pajak J, Jelonek M, Gasior P, Peppas A, Tellez A, Granada JF, Buszman PE. Experimental evaluation of pharmacokinetic profile and biological effect of a novel paclitaxel microcrystalline balloon coating in the iliofemoral territory of swine. Catheter Cardiovasc Interv. 2014 Feb;83(2):325-33. doi: 10.1002/ccd.24982. Epub 2013 Oct 23. PMID 23703720
- [Background] Tepe G, Zeller T, Albrecht T, Heller S, Schwarzwalder U, Beregi JP, Claussen CD, Oldenburg A, Scheller B, Speck U. Local delivery of paclitaxel to inhibit restenosis during angioplasty of the leg. N Engl J Med. 2008 Feb 14;358(7):689-99. doi: 10.1056/NEJMoa0706356. PMID 18272892
- [Background] Werk M, Langner S, Reinkensmeier B, Boettcher HF, Tepe G, Dietz U, Hosten N, Hamm B, Speck U, Ricke J. Inhibition of restenosis in femoropopliteal arteries: paclitaxel-coated versus uncoated balloon: femoral paclitaxel randomized pilot trial. Circulation. 2008 Sep 23;118(13):1358-65. doi: 10.1161/CIRCULATIONAHA.107.735985. Epub 2008 Sep 8. PMID 18779447
- [Background] Scheller B, Hehrlein C, Bocksch W, Rutsch W, Haghi D, Dietz U, Bohm M, Speck U. Treatment of coronary in-stent restenosis with a paclitaxel-coated balloon catheter. N Engl J Med. 2006 Nov 16;355(20):2113-24. doi: 10.1056/NEJMoa061254. Epub 2006 Nov 13. PMID 17101615
- [Background] Scheinert D, Duda S, Zeller T, Krankenberg H, Ricke J, Bosiers M, Tepe G, Naisbitt S, Rosenfield K. The LEVANT I (Lutonix paclitaxel-coated balloon for the prevention of femoropopliteal restenosis) trial for femoropopliteal revascularization: first-in-human randomized trial of low-dose drug-coated balloon versus uncoated balloon angioplasty. JACC Cardiovasc Interv. 2014 Jan;7(1):10-9. doi: 10.1016/j.jcin.2013.05.022. PMID 24456716
- [Derived] Nowakowski P, Uchto W, Hrycek E, Kachel M, Ludyga T, Polczyk F, Zurakowski A, Kazmierczak P, Granada JF, Nowakowska I, Kiesz RS, Milewski KP, Buszman PE, Buszman PP. Microcrystalline paclitaxel-coated balloon for revascularization of femoropopliteal artery disease: Three-year outcomes of the randomized BIOPAC trial. Vasc Med. 2021 Aug;26(4):401-408. doi: 10.1177/1358863X20988360. Epub 2021 Mar 9. PMID 33686879